CLINICAL TRIAL: NCT04535960
Title: Incretin and Treatment With Inhibition of Sodium-glucose Cotransporter-2 Combination Insights Into Mechanisms Implicated in Congestive Heart Failure: "NATRIURETIC" Trial
Acronym: NATRIURETIC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, David Z.I. Cherney, Associate Professor of Medicine, Clinician Scientist, University Health Network, Toronto
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 18-5058
Record Dates: First submitted 2020-02-12; First posted 2020-09-02 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: SGLT2 inhibition; GLP-1 receptor agonist; type 2 diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — empagliflozin; Liraglutide

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to initial therapy with empagliflozin 25mg PO daily or liraglutide 1.8 mg SC daily, for 6 weeks. After that, patients in the empagliflozin group will also receive liraglutide 1.8mg SC daily for additional 6 weeks and patients in the liraglutide group will also receive empagliflozin 25mg PO daily for 6 weeks (combination therapy).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Liraglutide (Experimental): Liraglutide Subcutaneous Total Dose 1.8mg daily for 6 weeks
  Interventions: Drug: Empagliflozin 25 MG + Liraglutide 1.8 MG; Drug: Liraglutide 1.8 MG + Empagliflozin 25 MG
- Empagliflozin (Experimental): Empagliflozin Tablets Total Dose 25mg daily for 6 weeks
  Interventions: Drug: Empagliflozin 25 MG + Liraglutide 1.8 MG; Drug: Liraglutide 1.8 MG + Empagliflozin 25 MG

INTERVENTIONS:
Drug: Empagliflozin 25 MG + Liraglutide 1.8 MG — Patients will be randomized to initial therapy with empagliflozin 25mg PO daily for 6 weeks. After that, patients in the empagliflozin group will also receive liraglutide 1.8mg SC daily for additional 6 weeks.
  Other Names: Generic names are above, listed
Drug: Liraglutide 1.8 MG + Empagliflozin 25 MG — Patients will be randomized to initial therapy with liraglutide 1.8 mg SC daily, for 6 weeks. After that, patients will also receive empagliflozin 25mg PO daily for 6 weeks.
  Other Names: Generic names are above, listed

SUMMARY:
This study aims to provide essential mechanistic insights into natriuretic and hemodynamic effects of SGLT2i and GLP-1RA agents in T2D patients. Ultimately, by obtaining physiological data in T2D patients without HF, our aims are to gain insight into how the use of this combined therapy may be used in T2D with HF in future work.

DETAILED DESCRIPTION:
Type 2 diabetes (T2D) is an epidemic that afflicts more than 350 million people world-wide. Despite the use of existing medical therapies, T2D continues to cause significant morbidity and mortality, leading to large societal and financial costs to Canadians.

Newer agents called sodium glucose co-transporter-2 inhibitors (SGLT2i) have been developed to improve glycemic control and lower hemoglobin A1c by increasing glycosuria. SGLT2i also reduce blood pressure and albuminuria in T2D - possibly through natriuresis. Importantly, a landmark trial "EMPA-REG OUTCOME" demonstrated that the SGLT2i empagliflozin is the first anti- hyperglycemic agent to reduce mortality and heart failure (HF) risk, and also to decrease the risk of progressive diabetic nephropathy.

Liraglutide, a glucagon-like peptide-1 receptor agonist (GLP-1RA), is a subcutaneous drug, used for treating T2D patients. Recently, this drug was also able to reduce cardiovascular endpoints in the LEADER trial. Furthermore, liraglutide attenuated the risk of progressive albuminuria as well. GLP-1RAs induce natriuretic effects, but have not been shown to reduce HF risk. Their positive cardiovascular effects are probably due to reduction in atherosclerotic events.

T2D patients are at high risk for development of both HF and atherosclerotic diseases. Given that SGLT2i and GLP-1RA seem to reduce cardiovascular outcomes via different approaches, combining these two agents in the treatment of T2D is an appealing new strategy. In this project, we aim to combine GLP-1RA and SGLT2i therapies in T2D patients without HF and compare renal and cardiovascular physiological measures in these patients, such as renal function, neurohormonal activation, blood pressure, arterial stiffness, and systemic vascular resistance. This could give a better understanding on the action of the combination therapy in T2D, support future mechanist trials with patients with HF, and give support to the development of large clinical trials on this topic.

Study design: Open-label, exploratory, randomized (with randomization concealment), pilot mechanistic trial, with two groups and 2 sequential treatments within each group.

Study population: Male and female subjects with T2D, 18 years old or older, with eGFR ≥30 mL/min/1.73m2, as described in the full protocol.

Intervention: Patients will be randomized to initial therapy with empagliflozin 25mg PO daily or liraglutide 1.8 mg SC daily, for 6 weeks. After that, patients in the empagliflozin group will also receive liraglutide 1.8mg SC daily for additional 6 weeks and patients in the liraglutide group will also receive empagliflozin 25mg PO daily for 6 weeks (combination therapy).

Primary Objective: Comparison of proximal tubular natriuresis (measured by FENa+, fractional excretion of sodium) after 6 weeks of SGLT2i monotherapy vs FENa+ after 6 weeks of combination therapy (SGLT2i + GLP-1RA) AND comparison of FENa+ after 6 weeks of GLP1-RA monotherapy vs FENa+ after 6 weeks of combination therapy (GLP-1RA + SGLT2i).

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Patients visit the outpatient clinic on a more regular basis than standard patient care - i.e. at study inclusion and at each study visit for clinical assessment. Blood work for physiological assessments, renal function tests and cardiovascular assessments will be obtained as described in the protocol. 24hr urine will be collected one day prior to the hospital visit. No other invasive measurements will be executed. Patients receive restitution of all travel costs and also a financial aid for 3 visits. Patients receive no priority in treatment of other diseases in the clinic during this study. There are no other direct benefits for the patients to be included and participation is on a voluntary basis.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women diagnosed with T2D ≥6 months prior to informed consent;
2. eGFR ≥30 mL/min/1.73m2;
3. Age >18 years;
4. HbA1c 7.0%-12.0%;
5. Body Mass Index (BMI) 18.5-40.0 kg/m2;
6. Stable HbA1c, measured 2-12 months prior to screening, within 5% of baseline value;
7. Blood pressure ≤160/100 mmHg at screening, >90/60 mmHg;
8. Stable on dose of ACE inhibitor, angiotensin receptor blocker or renin inhibitor for at least 2 weeks.

Exclusion Criteria:

1. Type 1 Diabetes;
2. Leukocyte and/or nitrite positive urinalysis that is untreated;
3. Severe hypoglycaemia within 2 months prior to screening;
4. History of hypoglycaemia unawareness based on investigator judgement;
5. Unstable coronary artery disease with acute coronary syndrome, percutaneous intervention or bypass surgery within 3 months;
6. Clinically significant valvular disease subject to PI/Sub PI's discretion;
7. Congestive heart failure subject to PI/Sub PI's discretion;
8. Bariatric surgery or other surgeries that induce chronic malabsorption within one year;
9. Anti-obesity drugs or diet regimen and unstable body weight three months prior to screening;
10. Treatment with systemic corticosteroids;
11. Blood dyscrasias or any disorders causing hemolysis or unstable red blood cells;
12. Pre-menopausal women who are nursing, pregnant, or of child-bearing potential and not practicing an acceptable method of birth control;
13. Participation in another trial with an investigational drug within 30 days of informed consent;
14. Alcohol or drug abuse within three months prior to informed consent that would interfere with trial participation or any ongoing clinical condition that would jeopardize subject safety or study compliance based on investigator judgement;
15. Liver disease, defined by serum levels of alanine transaminase, aspartate transaminase, or alkaline phosphatase >3 x upper limit of normal as determined during screening;
16. Medical history of cancer or treatment for cancer in the last five years prior to screening;
17. History of pancreatitis;
18. Personal of family history of medullary thyroid cancer or MEN2B;
19. Tachycardia, HR >100;
20. Use of SGLT2i, GLP-1RA or DPP-4i within the past 1 month (1-month minimum washout is allowed);
21. History of gastroparesis;
22. Known intolerance to SGLT2i or GLP-1RA;
23. Allergy to iodine-based substances if receiving iohexol for GFR measures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2019-01-24 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Proximal tubular natriuresis | up to 12 weeks
  Measured by fractional excretion of sodium

SECONDARY OUTCOMES:
Glomerular Filtration Rate | Glomerular Filtration Rate (GFR, based on plasma iohexol clearance) will be measured at 2 time points: monotherapy (6 weeks) and combination therapy (12 weeks)
  GFR
Systolic blood pressure | Systolic blood pressure (SBP) will be measured at 2 time points: monotherapy (6 weeks) and combination therapy (12 weeks)
  SBP
Body weight | Body weight will be measured at 2 time points: monotherapy (6 weeks) and combination therapy (12 weeks)
  Kilograms
Arterial stiffness | Arterial stiffness will be measured at 2 time points: monotherapy (6 weeks) and combination therapy (12 weeks)
  Measured using a Sphygmocor device
Systemic vascular resistance | Systemic vascular resistance will be measured at 2 time points: monotherapy (6 weeks) and combination therapy (12 weeks)
  Measured using non-invasive cardiac output monitor (NICOM)
Urinary concentration of the renin-angiotensin aldosterone system (RAAS) markers | Outcome will be measured at 2 time points: monotherapy (6 weeks) and combination therapy (12 weeks)
  Measured using ELISA
Urinary EGF,FGF2,Eotaxin,TGFa,G-CSF,Flt-3L,GM-CSF,Fractalkine,IFNa2,IFNy,GRO,IL10,MCP-3,IL-12P40,MDC,IL-12P70,PDGF-AA,IL-13,PDGF-BB,IL-15,sCD40L,IL-17A,IL-1RA,IL1a,IL9,IL1B,IL2,IL3,IL4,IL5,IL6,IL7,IL8,IL10,MCP-1,MIP-1a,MIP-1B,RANTES,TNFalpha,TNFB,VEGF | Outcome will be measured at 2 time points: monotherapy (6 weeks) and combination therapy (12 weeks)
  41-plex chemo/chemokine profile assay: urinary

CONTACTS AND LOCATIONS:
Overall Officials: David ZI Cherney, MD PhD FRCPC, Principal Investigator — University Health Network, Toronto General Hospital
Locations (1):
- Renal Physiology Laboratory, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No